CLINICAL TRIAL: NCT03325049
Title: The Health Promoting Conversations Intervention for Families With a Critically Ill Relative: A Pilot RCT
Brief Title: The Health Promoting Conversations for Families With a Critically Ill Relative
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We have closed the study because of slow inclusion of families
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Susanna Ågren, Head of the project, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LinkoepingU74
Record Dates: First submitted 2017-09-15; First posted 2017-10-30 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Family Health
Keywords: Family Relations; Family Health; Intervention study; Social support; Intensive care unit

STUDY DESIGN:
Intervention Model Description: This randomized controlled pilot study used a pre-test, post-test design with intervention and control groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The health-promoting conversations (Experimental): In the intervention group, there were 3 health-promoting conversations with each family after the discharge. The health-promoting conversations were held within an approximately 4- to 8-week period with an interval of 2 weeks between conversations. A closing letter was sent 2 to 3 weeks after the final conversation that summarized all of the conversations and that provided further opportunities for reflection.
  Interventions: Behavioral: The health-promoting conversations
- Control Arm (Active Comparator): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: The health-promoting conversations — The health-promoting conversations
  Arms: The health-promoting conversations
Other: Usual Care — Usual Care
  Arms: Control Arm

SUMMARY:
Objective: We investigated the outcomes of a nurse-led family intervention, Health Promoting Conversations, which focused on family functioning and wellbeing in families with a critically ill member.

Study design: This randomized controlled pilot study used a pre-test, post-test design with intervention and control groups to investigate the outcomes of the nurse-led intervention in 17 families.

Outcome measures: The Health Promoting Conversations intervention was evaluated using validated instruments that measure family functioning and family wellbeing: the General Functioning sub-scale from the McMaster Family Assessment Device; the Family Sense of Coherence, the Herth Hope Index, and the Medical Outcome Short-Form Health Survey. Descriptive and analytical statistical methods were used to analyse the data.

DETAILED DESCRIPTION:
This randomized control trial (RCT) used a pre-test, post-test design with intervention and control groups.

In the intervention group, there were 3 health-promoting conversations with each family after the discharge. The health-promoting conversations were held within an approximately 4- to 8-week period with an interval of 2 weeks between conversations. A closing letter was sent 2 to 3 weeks after the final conversation that summarized all of the conversations and that provided further opportunities for reflection.

Baseline data were collected to assess family functioning and wellbeing in the intervention group and the control group 1-2 months after the critical illness and before the start of the intervention. Follow-up assessments were conducted 3 and 12 months after the intervention for both groups. Additionally, background data, including health history, were collected using a self-administered questionnaire that asked about age; sex; education level; habits like smoking, alcohol consumption, and physical activity; psychosocial support; co-morbidity; and risk of mortality. The latter was calculated using the Charlson Comorbidity Index (Charlson et al., 1987).

The main outcome variables in this study were family functioning and family wellbeing. The following instruments were used in this study: 1) General Functioning (GF) sub-scale from the McMaster Family Assessment Device (FAD); 2) Family Sense of Coherence (F-SOC/F-KASAM); 3) Herth Hope Index (HHI); and 4) Medical Outcome Short-Form health survey (SF-36).

ELIGIBILITY:
Inclusion criteria:

* patient age >18 years
* patient treated in the ICU for at least 96 hours
* at least one family member (age >15 years) interested in participating

Exclusion criteria:

* dementia
* or other severe psychiatric illnesses
* drug abuse
* difficulties in understanding or reading the Swedish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
family functioning | up to 12 months
  e GF is a 12-item scale designed to measure self-reported perceived overall 15 family functioning (Wright and Leahey, 2009, 2013). Each item is rated on a four-point 16 Likert scale: 'strongly agree' = 1, 'agree' = 2, 'disagree' = 3 and 'strongly disagree' = 4. The 17 scale scores ranges from 12 to 48, with lower scores indicating better family functioning. The 18 GF was translated into Swedish and has been pilot tested in Swedish samples, and the scale 19 has shown satisfactory reliability and acceptable validity of 0.90 (Bylund et al., 2015). The 20 reliability coefficient alpha was 0.45 in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Ågren, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linköping university, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahlberg M, Backman C, Jones C, Walther S, Hollman Frisman G. Moving on in life after intensive care--partners' experience of group communication. Nurs Crit Care. 2015 Sep;20(5):256-63. doi: 10.1111/nicc.12192. Epub 2015 May 29. PMID 26032101
- [Background] Alderfer MA, Fiese BH, Gold JI, Cutuli JJ, Holmbeck GN, Goldbeck L, Chambers CT, Abad M, Spetter D, Patterson J. Evidence-based assessment in pediatric psychology: family measures. J Pediatr Psychol. 2008 Oct;33(9):1046-61; discussion 1062-4. doi: 10.1093/jpepsy/jsm083. Epub 2007 Sep 28. PMID 17905801
- [Background] Antonovsky, A., Sourani, T., 1988. Family sense of coherence and family adaption. Journal of Marriage and the Family. 50:79-92.
- [Background] Benzein E, Berg A. The Swedish version of Herth Hope Index--an instrument for palliative care. Scand J Caring Sci. 2003 Dec;17(4):409-15. doi: 10.1046/j.0283-9318.2003.00247.x. PMID 14629644
- [Background] Benzein EG, Hagberg M, Saveman BI. 'Being appropriately unusual': a challenge for nurses in health-promoting conversations with families. Nurs Inq. 2008 Jun;15(2):106-15. doi: 10.1111/j.1440-1800.2008.00401.x. PMID 18476853
- [Background] Benzein EG, Saveman BI. Health-promoting conversations about hope and suffering with couples in palliative care. Int J Palliat Nurs. 2008 Sep;14(9):439-45. doi: 10.12968/ijpn.2008.14.9.31124. PMID 19060795
- [Background] Benzein E, Olin C, Persson C. 'You put it all together' - families' evaluation of participating in Family Health Conversations. Scand J Caring Sci. 2015 Mar;29(1):136-44. doi: 10.1111/scs.12141. Epub 2014 Apr 9. PMID 24720612
- [Background] Bylund A, Arestedt K, Benzein E, Thorell A, Persson C. Assessment of family functioning: evaluation of the General Functioning Scale in a Swedish Bariatric Sample. Scand J Caring Sci. 2016 Sep;30(3):614-22. doi: 10.1111/scs.12269. Epub 2015 Nov 9. PMID 26555951
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Davydow DS, Gifford JM, Desai SV, Needham DM, Bienvenu OJ. Posttraumatic stress disorder in general intensive care unit survivors: a systematic review. Gen Hosp Psychiatry. 2008 Sep-Oct;30(5):421-34. doi: 10.1016/j.genhosppsych.2008.05.006. Epub 2008 Jul 30. PMID 18774425
- [Background] Dorell A, Isaksson U, Ostlund U, Sundin K. Family Health Conversations have Positive Outcomes on Families - A Mixed Method Research Study. Open Nurs J. 2017 Feb 28;11:14-25. doi: 10.2174/1874434601711010014. eCollection 2017. PMID 28400891
- [Background] Dowdy DW, Eid MP, Sedrakyan A, Mendez-Tellez PA, Pronovost PJ, Herridge MS, Needham DM. Quality of life in adult survivors of critical illness: a systematic review of the literature. Intensive Care Med. 2005 May;31(5):611-20. doi: 10.1007/s00134-005-2592-6. Epub 2005 Apr 1. PMID 15803303
- [Background] Dufault K, Martocchio BC. Symposium on compassionate care and the dying experience. Hope: its spheres and dimensions. Nurs Clin North Am. 1985 Jun;20(2):379-91. PMID 3846980
- [Background] Eggenberger SK, Nelms TP. Being family: the family experience when an adult member is hospitalized with a critical illness. J Clin Nurs. 2007 Sep;16(9):1618-28. doi: 10.1111/j.1365-2702.2007.01659.x. PMID 17727583
- [Background] Everson SA, Goldberg DE, Kaplan GA, Cohen RD, Pukkala E, Tuomilehto J, Salonen JT. Hopelessness and risk of mortality and incidence of myocardial infarction and cancer. Psychosom Med. 1996 Mar-Apr;58(2):113-21. doi: 10.1097/00006842-199603000-00003. PMID 8849626
- [Background] Everson SA, Kaplan GA, Goldberg DE, Salonen JT. Hypertension incidence is predicted by high levels of hopelessness in Finnish men. Hypertension. 2000 Feb;35(2):561-7. doi: 10.1161/01.hyp.35.2.561. PMID 10679498
- [Background] Frivold G, Slettebo A, Dale B. Family members' lived experiences of everyday life after intensive care treatment of a loved one: a phenomenological hermeneutical study. J Clin Nurs. 2016 Feb;25(3-4):392-402. doi: 10.1111/jocn.13059. PMID 26818366
- [Background] Fumis RR, Ranzani OT, Martins PS, Schettino G. Emotional disorders in pairs of patients and their family members during and after ICU stay. PLoS One. 2015 Jan 23;10(1):e0115332. doi: 10.1371/journal.pone.0115332. eCollection 2015. PMID 25616059
- [Background] Garvin P, Nilsson L, Carstensen J, Jonasson L, Kristenson M. Plasma levels of matrix metalloproteinase-9 are independently associated with psychosocial factors in a middle-aged normal population. Psychosom Med. 2009 Apr;71(3):292-300. doi: 10.1097/PSY.0b013e3181960e7f. Epub 2009 Feb 5. PMID 19196809
- [Background] Herth K. Abbreviated instrument to measure hope: development and psychometric evaluation. J Adv Nurs. 1992 Oct;17(10):1251-9. doi: 10.1111/j.1365-2648.1992.tb01843.x. PMID 1430629
- [Background] Jensen JF, Thomsen T, Overgaard D, Bestle MH, Christensen D, Egerod I. Erratum to: Impact of follow-up consultations for ICU survivors on post-ICU syndrome: a systematic review and meta-analysis. Intensive Care Med. 2015 Jul;41(7):1391. doi: 10.1007/s00134-015-3932-9. No abstract available. PMID 26104120
- [Background] Kose I, Zincircioglu C, Ozturk YK, Cakmak M, Guldogan EA, Demir HF, Senoglu N, Erbay RH, Gonullu M. Factors Affecting Anxiety and Depression Symptoms in Relatives of Intensive Care Unit Patients. J Intensive Care Med. 2016 Oct;31(9):611-7. doi: 10.1177/0885066615595791. Epub 2015 Jul 12. PMID 26168801
- [Background] Orwelius L, Kristenson M, Fredrikson M, Walther S, Sjoberg F. Hopelessness: Independent associations with health-related quality of life and short-term mortality after critical illness: A prospective, multicentre trial. J Crit Care. 2017 Oct;41:58-63. doi: 10.1016/j.jcrc.2017.04.044. Epub 2017 Apr 28. PMID 28482237
- [Background] Parker AM, Sricharoenchai T, Raparla S, Schneck KW, Bienvenu OJ, Needham DM. Posttraumatic stress disorder in critical illness survivors: a metaanalysis. Crit Care Med. 2015 May;43(5):1121-9. doi: 10.1097/CCM.0000000000000882. PMID 25654178
- [Background] Probst DR, Gustin JL, Goodman LF, Lorenz A, Wells-Di Gregorio SM. ICU versus Non-ICU Hospital Death: Family Member Complicated Grief, Posttraumatic Stress, and Depressive Symptoms. J Palliat Med. 2016 Apr;19(4):387-93. doi: 10.1089/jpm.2015.0120. Epub 2016 Feb 1. PMID 26828564
- [Background] Ridenour TA, Daley JG, Reich W. Factor analyses of the family assessment device. Fam Process. 1999 Winter;38(4):497-510. doi: 10.1111/j.1545-5300.1999.00497.x. PMID 10668625
- [Background] Sagy S, Dotan N. Coping resources of maltreated children in the family: a salutogenic approach. Child Abuse Negl. 2001 Nov;25(11):1463-80. doi: 10.1016/s0145-2134(01)00285-x. PMID 11766011
- [Background] Svenningsen H, Langhorn L, Agard AS, Dreyer P. Post-ICU symptoms, consequences, and follow-up: an integrative review. Nurs Crit Care. 2017 Jul;22(4):212-220. doi: 10.1111/nicc.12165. Epub 2015 Feb 17. PMID 25688675
- [Background] Tilburgs B, Nijkamp MD, Bakker EC, van der Hoeven H. The influence of social support on patients' quality of life after an intensive care unit discharge: A cross-sectional survey. Intensive Crit Care Nurs. 2015 Dec;31(6):336-42. doi: 10.1016/j.iccn.2015.07.002. Epub 2015 Aug 28. PMID 26321655
- [Background] Ullman AJ, Aitken LM, Rattray J, Kenardy J, Le Brocque R, MacGillivray S, Hull AM. Intensive care diaries to promote recovery for patients and families after critical illness: A Cochrane Systematic Review. Int J Nurs Stud. 2015 Jul;52(7):1243-53. doi: 10.1016/j.ijnurstu.2015.03.020. Epub 2015 Apr 4. PMID 25869586
- [Background] van Beusekom I, Bakhshi-Raiez F, de Keizer NF, Dongelmans DA, van der Schaaf M. Reported burden on informal caregivers of ICU survivors: a literature review. Crit Care. 2016 Jan 21;20:16. doi: 10.1186/s13054-016-1185-9. PMID 26792081
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Ware, JE., 1993. SF-36 health survey manual and interpretation guide., Boston., The New Health Institute, New England Medical Center.
- [Background] Ware, J., Kosinski, M., Dewey, J., 2001. How to score version 2 of the SF-36 health survey. In.Rhode Island, USA: Quality Metric Incorporated; Lincoln.
- [Background] WMA, The World Medical Association., 2013. Declaration of Helsinki - Etical Principals for 10 Medical Research Involving Human Subjects, 11 https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-12 medical-research-involving-human-subjects/
- [Background] Wright, LM., Leahey, M., 2009. Nurses and families: A guide to family assessment and 14 intervention (5 Rev ed ed.). Pennsylvania: F.A. Davis Company.
- [Background] Wright, LM., Leahey, M., 2013. Nurses and families: A guide to family assessment and 17 intervention (6th ed.). Philadelphia, PA: F.A. Davis.
- [Background] Wahlin I, Ek AC, Idvall E. Patient empowerment in intensive care--an interview study. Intensive Crit Care Nurs. 2006 Dec;22(6):370-7. doi: 10.1016/j.iccn.2006.05.003. Epub 2006 Aug 4. PMID 16890438
- [Background] Agard AS, Egerod I, Tonnesen E, Lomborg K. From spouse to caregiver and back: a grounded theory study of post-intensive care unit spousal caregiving. J Adv Nurs. 2015 Aug;71(8):1892-903. doi: 10.1111/jan.12657. Epub 2015 Apr 1. PMID 25827018